CLINICAL TRIAL: NCT03815864
Title: Role of Donor Specific Antibodies, Other Anti-human Leucocyte Antibodies and Autoantibodies in the Outcome of Liver Retransplantation
Brief Title: Antibodies and Liver Retransplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Vivian McAlister, Professor of Surgery, London Health Sciences Centre
Other Study IDs: 106961
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Liver Transplant Failure; Antibody-mediated Rejection
Keywords: donor specific antibody; autoantibody; human leucocyte antigen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples stored for clinical use by the Transplant Laboratory since the beginning of liver transplantation at our facility in 1977
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D2SA+: Median fluoresce intensity > or = 1000 on Luminex-based solid phase assay of banked sera for anti-HLA antibodies directed against the donor of a second liver transplantation
  Interventions: Diagnostic Test: Luminex-based solid phase assay of banked sera for anti-HLA antibodies directed against the donor of a second liver transplantation
- D2SA-: Median fluoresce intensity < 1000 on Luminex-based solid phase assay of banked sera for anti-HLA antibodies directed against the donor of a second liver transplantation
  Interventions: Diagnostic Test: Luminex-based solid phase assay of banked sera for anti-HLA antibodies directed against the donor of a second liver transplantation

INTERVENTIONS:
Diagnostic Test: Luminex-based solid phase assay of banked sera for anti-HLA antibodies directed against the donor of a second liver transplantation — Anti-AT1R antibodies were tested on pre-transplantation sera using ELISA kit (Lot #30, One Lambda, Canoga Park, CA)
  Other Names: AT1R antibody

SUMMARY:
Despite reports that associate donor specific antibody (DSA) with rejection after liver transplantation, grafts are still allocated according to blood group (ABO) but not human leukocyte antigen (HLA) compatibility, possibly due to the absence of an easily discernible clinical association between adverse recipient outcome and DSA. Re-transplantation provides a test environment where the presence of preformed DSA or other antibodies is prevalent and events (graft loss) more common so that the effect of these antibodies on outcome should be apparent. This is an observational study of routine clinical care to determine these effects on our own patients. The goal is to perfect donor-recipient matching to attain the best outcome. In addition, we may develop hypotheses and potential treatments that would be tested in further clinical trials

DETAILED DESCRIPTION:
Despite reports that associate donor specific antibody (DSA) with rejection after liver transplantation, grafts are still allocated according to blood group (ABO) but not human leukocyte antigen (HLA) compatibility, possibly due to the absence of an easily discernible clinical association between adverse recipient outcome and DSA. Re-transplantation provides a test environment where the presence of preformed DSA or other antibodies is prevalent and events (graft loss) more common so that the effect of these antibodies on outcome should be apparent. This is an observational study of routine clinical care to determine these effects on our own patients.

In phase 1, we will examine the effect of antibodies specifically directed against the second donor in liver retransplantation. Other factors known to effect the outcome will be checked to allow for risk adjustment.

In phase 2, we will examine the role played by specific auto-antibodies such as angiotensin II receptor type 1 antibodies and endothelin-1 type A receptor antibodies on the outcome of liver retransplantation.

The goal of these observational study is to perfect donor-recipient matching to attain the best outcome. In addition, we may develop hypotheses and potential treatments that would be tested in further clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a second liver transplantation performed at LHSC

Exclusion Criteria:

* Recipients of ABO incompatible second liver transplantation
* Recipients of multiple organs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients who have undergone a repeat transplantation of the liver at LHSC.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 1977-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Retransplant graft survival | From date of transplantation until the date of next transplantation or date of death from any cause, whichever came first, assessed up to 240 months
  Average length of time the second liver graft remains in a living recipient regardless of function

SECONDARY OUTCOMES:
Patient survival | From date of transplantation until the date of death from any cause assessed up to 240 months
  Average length of time a recipient is alive regardless of presence of the second liver transplant

OTHER OUTCOMES:
Acute rejection | From date of transplantation until the date of first documented acute rejection assessed up to 240 months
  number of participants with a clinically diagnosed and treated episode of rejection (either acute cellular or humoral)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian McAlister, Principal Investigator — London Health Sciences Center

IPD SHARING:
Plan to Share IPD: Yes
Study mechanisms and de-identified subject level data will be shared with researchers who contact the principal investigator.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: From publication until 5 years later
Access Criteria: De-identified subject level data will be shared with researchers who contact the principal investigator, submit a research plan and sign an agreement. Approval by Western Research Ethics may be required depending on the request.

REFERENCES:
- [Derived] Xu Q, McAlister VC, House AA, Molinari M, Leckie S, Zeevi A. Autoantibodies to LG3 are associated with poor long-term survival after liver retransplantation. Clin Transplant. 2021 Jul;35(7):e14318. doi: 10.1111/ctr.14318. Epub 2021 Apr 25. PMID 33871888
- [Derived] Xu Q, McAlister VC, Leckie S, House AA, Skaro A, Marotta P. Angiotensin II type I receptor agonistic autoantibodies are associated with poor allograft survival in liver retransplantation. Am J Transplant. 2020 Jan;20(1):282-288. doi: 10.1111/ajt.15571. Epub 2019 Sep 6. PMID 31419065